CLINICAL TRIAL: NCT01089023
Title: Multicenter, Open-Label Study to Evaluate the Safety, Tolerability and the Effect on Disease Activity of Tocilizumab in Patients With Active Rheumatoid Arthritis on Background Non-biologic DMARDs Who Have an Inadequate Response to Current Non-biologic DMARD and/or Anti- TNF Therapy.
Brief Title: A Study of Tocilizumab as Monotherapy or in Combination With DMARDs in Patients With Moderate to Severe Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22440
Record Dates: First submitted 2010-03-08; First posted 2010-03-18 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg iv infusion, every 4 weeks for a total of 6 infusions

SUMMARY:
This open-label single-arm study will evaluate the safety, tolerability and efficacy of tocilizumab [RoActemra/Actemra] in patients with moderate to severe rheumatoid arthritis who experience an inadequate clinical response to a stable dose of non-biologic disease modifying anti-rheumatic drugs (DMARD) or anti-tumor necrosis factors (TNFs). RoActemra/Actemra will be administered as a monotherapy or in combination with DMARDs. RoActemra/Actemra will be administered as intravenous infusion at a dose of 8 mg/kg every 4 weeks for a total of 6 infusions. The anticipated time on study treatment is 24 weeks. The target sample size is 50-150 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/=18 years of age
* moderate to severe rheumatoid arthritis (DAS28 >3.2) of 6 months duration
* inadequate clinical response to non-biologic DMARDs or anti-TNF
* bodyweight </=150 kg

Exclusion Criteria:

* rheumatic autoimmune disease or inflammatory joint disease other than RA
* major surgery within 8 weeks prior to screening or planned major surgery within 6 months following screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Bahrain (2):
  - Manama
  - Riffa
- Iran (2):
  - Isfahan
  - Tehran
- Safat, Kuwait
- Doha, Qatar
- Abu Dhabi, United Arab Emirates

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab 8 Milligrams Per Kilogram (mg/kg): Participants received tocilizumab 8 mg/kg intravenous (IV) infusion, once every 4 weeks for a total of 6 infusions.
Period: Overall Study
Arm/Group | Tocilizumab 8 Milligrams Per Kilogram (mg/kg)
Started | 95
Completed | 88
Not Completed | 7
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: All the participants who were administered treatment at each visit were considered during the analysis.
Groups:
- Tocilizumab 8 mg/kg: Participants received tocilizumab 8 mg/kg IV infusion, once every 4 weeks for a total of 6 infusions.
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.89 (13.677)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Any Adverse Event - Overall Summary of Events
Description: Percentage of participants with a serious adverse event (SAE), who died, with an adverse event (AE), or study drug related AE during the study.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, and 24
Population: All the participants who were administered treatment at each visit were considered during the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 95
percentage of participants
  With an SAE | 8.4
  Who Died | 0
  With any drug-related AE | 38.9
  With any AE | 45.3

2. Secondary Outcome: Percentage of Participants by Disease Activity Score Based on 28-Joint Count (DAS28) Category
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]) and global health assessment (participant rated global assessment of disease activity using 10-mm Visual analog scale - VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. A DAS28 score of greater than (>)5.1 indicated high disease activity, a score of >3.2 but less than or equal to (≤)5.1 indicated moderate disease activity, a score of greater than or equal to (≥)2.6 but ≤3.2 indicated low disease activity, and a score of less than <2.6 indicated disease remission. Week 24 is the Follow-Up visit.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: All the participants who were administered treatment at each visit were considered during the analysis.
  n (number) at Week 24 equals (=) number of participants in that visit; n at Other Visits = number of participants with treatment administered
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 95
percentage of participants
  High Disease Activity, Baseline (n=95) | 66.3
  High Disease Activity, Week 4 (n=93) | 15.1
  High Disease Activity, Week 8 (n=91) | 5.5
  High Disease Activity, Week 12 (n=89) | 2.2
  High Disease Activity, Week 16 (n=89) | 3.4
  High Disease Activity, Week 20 (n=88) | 1.1
  High Disease Activity, Week 24 (n=95) | 0
  Moderate Disease Activity, Baseline (n=95) | 33.7
  Moderate Disease Activity, Week 4 (n=93) | 48.4
  Moderate Disease Activity, Week 8 (n=91) | 36.3
  Moderate Disease Activity, Week 12 (n=89) | 23.6
  Moderate Disease Activity, Week 16 (n=89) | 11.2
  Moderate Disease Activity, Week 20 (n=88) | 10.2
  Moderate Disease Activity, Week 24 (n=95) | 7.4
  Low Disease Activity, Baseline (n=95) | 0.0
  Low Disease Activity, Week 4 (n=93) | 26.9
  Low Disease Activity, Week 8 (n=91) | 26.4
  Low Disease Activity, Week 12 (n=89) | 36.0
  Low Disease Activity, Week 16 (n=89) | 16.9
  Low Disease Activity Week 20 (n=88) | 15.9
  Low Disease Activity Week 24 (n=95) | 23.2
  Remission Baseline (n=95) | 0
  Remission Week 4 (n=93) | 9.7
  Remission Week 8 (n=91) | 31.9
  Remission Week 12 (n=89) | 38.2
  Remission Week 16 (n=89) | 67.4
  Remission Week 20 (n=88) | 67.4
  Remission Week 24 (n=95) | 64.2

3. Secondary Outcome: Percentage of Participants Achieving a Clinically Meaningful Improvement as Measured by DAS28
Description: DAS28 was calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hr) and global health assessment (participant rated global assessment of disease activity using 10-mm VAS); DAS28 score ranged from 0 to 10, where higher scores correspond to greater disease activity. Participants achieved a clinically meaningful improvement in DAS28 if there was a reduction of at least 1.2 units from baseline.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: All the participants who were administered treatment at each visit were considered during the analysis.
  n at Week 24 = number of participants in that visit; n at Other Visits = number of participants with treatment administered
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 95
percentage of participants
  Week 4 (n=93) | 82.8
  Week 8 (n=91) | 92.3
  Week 12 (n=89) | 95.5
  Week 16 (n=89) | 95.5
  Week 20 (n=88) | 94.3
  Week 24 (n=95) | 91.6

4. Secondary Outcome: Time to DAS28 Response by DAS28 Category
Description: Time to response is the number of days from date of first infusion to date of event. DAS28 response was defined as achievement of Low Disease Activity (DAS28 ≥2.6 to ≤3.2), Remission (DAS28 <2.6), or Clinically Meaningful Improvement (change of >1.2 from baseline).
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: All the participants who were administered treatment at each visit were considered during the analysis.
Measure: Mean (Standard Error); unit: days
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 95
days
  Clinically meaningful Improvement in DAS28 | 36.430 (2.355)
  Low disease activity (≥2.6 to ≤3.2) | 75.261 (5.587)
  Remission (<2.6) | 89.945 (4.395)

5. Secondary Outcome: Percentage of Participants With a Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) of at Least 0.22 Units
Description: HAQ includes 20 questions concerning participant's activities of daily life, grouped in 8 scales of 2 to 3 questions for each activity. To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Scoring was as follows with respect to performance of participant's everyday activities: 0=without difficulties; 1= with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. Minimum score was 0, maximum score was 3.
Time Frame: Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 95
percentage of participants
  Week 4 (n=93) | 61.3
  Week 8 (n=91) | 72.5
  Week 12 (n=89) | 87.6
  Week 16 (n=89) | 93.3
  Week 20 (n=88) | 92.0
  Week 24 (n=95) | 83.2

6. Secondary Outcome: Percentage of Participants With Improvement in Physical Function by HAQ-DI Category
Description: Physical function scoring was as follows with respect to performance of participant's everyday activities: 0=without difficulties; 1= with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. Minimum score was 0, maximum score was 3. The HAQ-DI score at every visit was categorized into none to mild disability (HAQ-DI <1), moderate disability (1≤ HAQ-DI <2) and severe disability (HAQ-DI ≥2). The percentages of the participants falling in each of these categories with respect to the visits were determined.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 95
percentage of participants
  HAQ-DI <1 Baseline (n=95) | 13.7
  HAQ-DI <1 Week 4 (n=93) | 36.6
  HAQ-DI <1 Week 8 (n=91) | 50.5
  HAQ-DI <1 Week 12 (n=89) | 60.7
  HAQ-DI <1 Week 16 (n=89) | 73.0
  HAQ-DI <1 Week 20 (n=88) | 80.7
  HAQ-DI <1 Week 24 (n=95) | 71.6
  ≤1 HAQ-DI <2 Baseline (n=95) | 61.1
  ≤1 HAQ-DI <2 Week 4 (n=93) | 46.2
  ≤1 HAQ-DI <2 Week 8 (n=91) | 39.6
  ≤1 HAQ-DI <2 Week 12 (n=89) | 34.8
  ≤1 HAQ-DI <2 Week 16 (n=89) | 25.8
  ≤1 HAQ-DI <2 Week 20 (n=88) | 15.9
  ≤1 HAQ-DI <2 Week 24 (n=95) | 15.8
  HAQ-DI ≥2 Baseline (n=95) | 24.2
  HAQ-DI ≥2 Week 4 (n=93) | 17.2
  HAQ-DI ≥2 Week 8 (n=91) | 9.9
  HAQ-DI ≥2 Week 12 (n=89) | 4.5
  HAQ-DI ≥2 Week 16 (n=89) | 1.1
  HAQ-DI ≥2 Week 20 (n=88) | 2.3
  HAQ-DI ≥2 Week 24 (n=95) | 3.2

7. Secondary Outcome: HAQ-DI Score by Visit
Description: as for outcome 5
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 95
scores on a scale
  Baseline (n=95) | 1.570 (0.6157)
  Week 4 (n=93) | 1.185 (0.7092)
  Week 8 (n=91) | 0.972 (0.6236)
  Week 12 (n=89) | 0.805 (0.5634)
  Week 16 (n=89) | 0.680 (0.4804)
  Week 20 (n=88) | 0.576 (0.4812)
  Week 24 (n=95) | 0.551 (0.5139)

8. Secondary Outcome: C-Reactive Protein (CRP) Values by Study Visit
Description: CRP is an acute phase inflammatory marker. The serum concentration of CRP is measured in milligrams per liter (mg/L). A reduction in the level is considered an improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: All the participants who were administered treatment at each visit were considered during the analysis.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 95
mg/L
  Baseline | 26.90 (34.406)
  Week 4 | 8.49 (29.074)
  Week 8 | 7.84 (23.116)
  Week 12 | 5.32 (10.614)
  Week 16 | 5.18 (8.105)
  Week 20 | 5.62 (8.618)
  Week 24 | 8.59 (21.702)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Test type: Superiority or Other; p < 0.0001, ANOVA — p-value measures the significance between each visit using analysis of variance

9. Secondary Outcome: Erythrocyte Sedimentation Rate
Description: ESR (measured in mm/hr) is an inflammation marker used to determine acute phase response.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20, and 24
Population: All the participants who were administered treatment at each visit were considered during the analysis.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab 8 mg/kg
Number analyzed (Participants) | 95
mm/hr
  Baseline | 45.27 (29.227)
  Week 4 | 10.61 (14.118)
  Week 8 | 7.66 (11.554)
  Week 12 | 7.52 (10.361)
  Week 16 | 5.83 (6.386)
  Week 20 | 6.60 (8.576)
  Week 24 | 9.17 (12.311)
Statistical Analysis 1: Comparison: Tocilizumab 8 mg/kg; Test type: Superiority or Other; p < 0.0001, ANOVA — p-value measures the significance between each visit using analysis of variance

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the date of first dose of study drug administration to the end of study at Week 24.
Description: Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events. Note that available data included a summary of events by system organ class only, no data provided by preferred term.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg iv infusion, every 4 weeks for a total of 6 infusions.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 8/95
Other Adverse Events (participants affected / at risk) | 43/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=95)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 3
Investigations (Investigations) | 2
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2
Infection and infestation (Infections and infestations) | 1
Renal and urinary disorders (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=95)
Investigations (Investigations) | 29
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 7
Infections and infestations (Infections and infestations) | 7
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 7
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 5
Gastrointestinal disorders (Gastrointestinal disorders) | 4
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 4
General disorders and administration site conditions (General disorders) | 3
Nervous system disorders (Nervous system disorders) | 3
Respiratory, thoracic, and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3
Cardiac disorders (Cardiac disorders) | 1
Injury, poisoning, and procedural complications (Injury, poisoning and procedural complications) | 1
Renal and urinary disorders (Renal and urinary disorders) | 1
Vascular disorders (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.